CLINICAL TRIAL: NCT01547364
Title: Blinded Analgesic Effect and 1 Year Outcome of Caudal D5W Injection in All-Comers With Chronic Low Back Pain and Either Buttock or Leg Pain
Brief Title: Caudal Epidural Injection of Dextrose For Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Smigel, Liza, M.D. (Individual)
Responsible Party: Principal Investigator, Liza Smigel, M.D., Liza Smigel, M.D., Smigel, Liza, M.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SweetCaudal
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Caudal; Epidural; Dextrose; Analgesia; TRVP1
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride; Saline Solution; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caudal Saline (Placebo Comparator)
  Interventions: Drug: Saline
- Caudal Dextrose (Active Comparator)
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Saline — Injection of 10 ml of normal saline into the caudal epidural space
  Other Names: Normal Saline
  Arms: Caudal Saline
Drug: Dextrose — Injection of 10 ml or dextrose 5% in water into the caudal epidural space
  Other Names: D5W
  Arms: Caudal Dextrose

SUMMARY:
Objective: The purposes of the study are to

1. Explore the immediate and short term (to 48 hour) analgesic potential of epidural D5W in comparison to normal saline.
2. Determine if cumulative benefit results from caudal dextrose injection.
3. Evaluate accuracy of a small needle vertical approach caudal injection that will allow for blind injection of D5W.

DETAILED DESCRIPTION:
Injection of dextrose into the epidural space as an admixture with various steroids and anesthetic has been utilized for years for purposes of altering the specific gravity of the injectate. No safety issues or concerns have been raised about the dextrose component inclusion but a separate therapeutic effect of dextrose has not heretofore been considered. Recently dextrose has been found to treat neurogenic inflammation (pain from upregulation of the TRPV1 receptor on peptidergic nerves). An analgesic effect of dextrose on chronic pain in the presence of painful sensory nerves has been observed with injection of D5W without anesthetic. That effect begins within seconds clinically. Physicians have empirically trialed D5W for epidural injection in a 10 ml volume and found that marked or complete analgesia of chronic low back and leg pain results in the majority of patients within 15 minutes. An empirical consecutive patient date collection has demonstrated that this initial effect lasts for 2 to 48 hours, and that the effect begins to sustain after 2-3 sessions. For this reason, the current study is designed with the the first two objectives:

1. Explore the immediate and short term (to 48 hour) analgesic potential of epidural D5W in comparison to normal saline.
2. Determine if cumulative benefit results from caudal dextrose injection.

In addition to determining potential benefit from caudal epidural of dextrose, the accuracy of a simple vertical approach to injection of dextrose is to be evaluated. If this vertical approach is accurate it will allow for

1. More comfort with injection.
2. Less need for radiographic exposure, in that needle placement is quicker and easier, allowing for less fluoroscopy time.
3. Potential for blind injection of solutions that do not include anesthetic or particulate matter, increasing potential applicability of caudal dextrose injection to situations in which fluoroscopy is not available.

ELIGIBILITY:
Inclusion Criteria:

* More than 3 months of back pain
* Some pain below the iliac crest (Either in buttock or in leg)
* At least one conservative (non-injection) modality of treatment to include physical therapy, chiropractic/osteopathic manipulation, exercises, drug therapy, and relative rest.
* Opiate use absent or controlled
* Psychiatric history absent or controlled
* Current medical stability
* Absent steroid use history or no allergy or intolerance to steroid use

Exclusion Criteria:

* Unstable neurologic function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 20 minutes in Numerical Rating Scale(NRS) for Pain | 20 minutes
  Caudal epidural injection of D5W will result in more analgesia at 20 minutes than epidural injection of normal saline.

SECONDARY OUTCOMES:
Change from Baseline to 1 year in NRS for Pain | 1 year
  Those with consistent analgesia after caudal epidural dextrose will note cumulative benefit on pain and disability that will exceed 1.5 times the MCID for pain and disability in low back pain. (NRS change of 3 or more)
Percentage Success of Epidurogram Pattern Production with a Blind Needle Placement Using a Vertical Caudal Epidural Method | Dye instillation immediately after needle placement with observation of dye pattern fluoroscopically.
  Blind use of the Rosen technique for vertical short needle caudal epidural injection will produce an epidurogram pattern 80% of the time upon first needle placement.

CONTACTS AND LOCATIONS:
Overall Officials: Liza Smigel, M.D., Principal Investigator — Liza Smigel, M.D., P.A.
Locations (1):
- Liza Smigel, M.D., Hilo, Hawaii, United States